CLINICAL TRIAL: NCT03950401
Title: Prospective Randomized Trial of Monocryl Versus Nylon Suture Closure in Carpal Tunnel Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1386423
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: skin closure
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — glycolide E-caprolactone copolymer; Nylons

STUDY DESIGN:
Intervention Model Description: Randomization to Monocryl versus subcuticular Nylon type of skin closure.
Who Masked: Outcomes Assessor
Masking Description: There is no way to mask the two techniques from the provider or patient since they will see the final result of the technique. The data analysis can be performed in a blinded manner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Monocryl (Active Comparator): Closure of the skin at the completion of surgery by interrupted subcuticular technique with absorbable Monocryl suture.
  Interventions: Procedure: Monocryl
- Nylon (Active Comparator): Closure of the skin at the completion of surgery by interrupted technique on top of the skin with non-absorbable Nylon suture. These will be removed at the first postoperative visit.
  Interventions: Procedure: Nylon

INTERVENTIONS:
Procedure: Monocryl — subcuticular Monocryl wound closure
  Arms: Monocryl
Procedure: Nylon — wound closure using nylon suture on the skin
  Arms: Nylon

SUMMARY:
The investigators will compare the early postoperative outcome of wound closure technique in carpal tunnel release using Nylon sutures versus subcuticular Monocryl sutures. The investigators plan to randomize patients across three hand surgeons who will perform both techniques, and will survey the patients satisfaction of pain and appearance at 2 and 6 weeks postoperatively.

DETAILED DESCRIPTION:
Objectives:

The aim of this study is to determine if there is a significant difference in provider-assessed and patient-assessed outcomes using subcuticular Monocryl vs traditional Nylon sutures for wound closure following open carpal tunnel decompression surgery.

Null hypothesis: There is no significant difference in provider-assessed or patient-assessed outcomes, as measured by the Patient and Observer Scar Assessment Scale (POSAS), between subcuticular Monocryl and traditional nylon wound closure methods after open carpal tunnel surgery.

Alternative hypothesis: Using a running subcuticular Monocryl suture for wound closure following open carpal tunnel release will result in significantly improved POSAS scores in comparison to traditional nylon wound closure

Background:

Open carpal tunnel decompression surgery is a common procedure, but controversy still exists regarding what wound closure method optimizes wound healing, cosmetic and patient satisfaction outcomes.

Research concerning the superiority of absorbable or non-absorbable sutures in the setting of wound closure for carpal tunnel decompression surgery is largely inconclusive, due to high risk of bias in previous comparison trials. Although some studies suggest that absorbable sutures confer a higher risk of infection, other studies suggest that absorbable sutures confer superior pain reduction, and still others suggest use of non-absorbable sutures due to reduced cost, both with respect to materials and by avoiding an additional clinician visit for suture removal.

A rigorous randomized trial of absorbable versus non-absorbable sutures as wound closure methods following minor elective hand surgery procedures is indicated, to compare wound healing, cosmesis, patient-reported outcome measures, as well as cost for each method.

Study Timelines:

Participants will be enrolled either at their pre-operative clinic visit or on the day of their surgery in the preoperative holding area (PHA). They will receive 2 follow-up appointments at 10-14 days and 6 weeks, after the surgery. Patients are considered enrolled in the study until after their 6-week appointment.

Power Analysis:

The power analysis will use alpha = 0.05 and beta (power) = 0.8. Using the Fleisher et al. paper, the mean Observer Scar Assessment Scale (OSAS) was 12 ± 3 for the suture group (p < 0.01), and the mean for the staple group was 13. If the investigators expect to see a similar difference between absorbable versus non-absorbable sutures, based on a two-sample t-test they would have to enroll 141 patients in each arm to have an 80% chance of seeing a difference at least this large, if there truly is one.

It is anticipated that a small percentage of patients will drop out of the study prior to completing their study endpoints. If the study allows for an approximate 15% dropout rate, then the investigators will plan to enroll 325 patients to ensure appropriate power. Looking at the surgeon numbers, each of the primary surgeons perform between 50-90 carpal tunnel surgeries per year. Therefore, the investigators estimate a 2.5 year enrollment period, followed by a six-month data review period.

Study Endpoints:

The primary study endpoint for subjects is a completed POSAS surveys at 6 weeks after their surgery.

There are no safety endpoints, as the study consists of a single intervention and both closure methods are well described and well tolerated (non-experimental).

Procedures Involved:

Patients will be identified by the operating surgeon (Dr. Szabo, Dr. Bayne or Dr. Allen) and enrolled either at their pre-operative clinic visit or in the preoperative holding area on the day of their surgery by either the operating surgeon or research personnel. After signing consent, the consenting researcher will use a digital Randomizer application ("Randomizer", available on all smart phones) to assign the individual to either Subcuticular Monocryl wound closure or traditional nylon wound closure. After being randomized, the study arm will be noted at the top of their consents and the consent scanned into the patient's electronic medical record. The hard copy consents will be stored securely as outlined below.

Patients will undergo surgery with the assigned wound closure. At each follow-up appointment (at approximately 2 and 6 weeks), patients and their operating physician will be given the POSAS questionnaire. In addition, patients will be asked the following question: "How satisfied are you with the results of the carpal tunnel surgery and recovery?" Assessed using a 5-point scale: completely satisfied (1 point), very satisfied (2 point), rather satisfied (3 point), dissatisfied (4 point), and completely dissatisfied (5 point).

Outcomes of the POSAS and satisfaction question will be complied into a research database and the de-identified data will be analyzed for significant differences between Subcuticular Monocryl and traditional nylon methods of wound closure.

During the data analysis phase of the study, a cost comparison will be performed, examining the cost of materials for each arm (assuming one suture packet used per patient). The investigators will also consider the cost differential in follow up visits, if patients closed with absorbable Monocryl sutures could be limited to one 6-week follow up visit, versus the nylon closure patients which would need an additional early visit for suture removal. No protected health information will need to be examined for this analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the University of California, Davis Health Center who are scheduled to undergo surgery for carpal tunnel release will be screened for eligibility for this study.
* Patients who do not speak English will be included in this study, and will be provided with appropriate translators at all communication points.

Exclusion Criteria:

* Patients who are not able to follow up at the 2 and 6 week postoperative time points.
* Patients who have known skin sensitivity to tape or absorbable suture.
* Those who are unable to give informed consent, individuals who are not yet adults (18 years or older), pregnant women, and prisoners will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) Score - Patient | 6 weeks
  As measured by a questionnaire completed by the patient. The patient scale consists of 6 items scored on a scale ranging from 1 ('no, not at all' or 'no, normal skin') to 10 ('yes, very much' or 'yes, very different'). Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.
Patient and Observer Scar Assessment Scale (POSAS) Score - Observer | 6 weeks
  As measured by a questionnaire completed by the clinic physician assistant. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area). All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks
  Patients will be asked the following question: "How satisfied are you with the results of the carpal tunnel surgery and recovery?" Assessed using a 5-point scale: completely satisfied (1 point), very satisfied (2 point), rather satisfied (3 point), dissatisfied (4 point), and completely dissatisfied (5 point).

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Szabo, MD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Correspondence of participants, their status in the study and the survey questions will be through encrypted excel document within encrypted OneDrive sharing folder with a link that is personally sent to the participants of the study.
Supporting Information: Study Protocol, ICF
Time Frame: Upon first patient enrollment, until completion of data analysis, likely at 2 years.
Access Criteria: Completed HIPAA and human subjects research training as enforced by University of California, Davis, and included as a participant of the study.

REFERENCES:
- [Background] Wade RG, Wormald JC, Figus A. Absorbable versus non-absorbable sutures for skin closure after carpal tunnel decompression surgery. Cochrane Database Syst Rev. 2018 Feb 1;2(2):CD011757. doi: 10.1002/14651858.CD011757.pub2. PMID 29390170
- [Background] Menovsky T, Bartels RH, van Lindert EL, Grotenhuis JA. Skin closure in carpal tunnel surgery: a prospective comparative study between nylon, polyglactin 910 and stainless steel sutures. Hand Surg. 2004 Jul;9(1):35-8. doi: 10.1142/s0218810404002017. PMID 15368623
- [Background] Hansen TB, Kirkeby L, Fisker H, Larsen K. Randomised controlled study of two different techniques of skin suture in endoscopic release of carpal tunnel. Scand J Plast Reconstr Surg Hand Surg. 2009;43(6):335-8. doi: 10.1080/02844310902955763. PMID 19995253
- [Background] Fleisher J, Khalifeh A, Pettker C, Berghella V, Dabbish N, Mackeen AD. Patient satisfaction and cosmetic outcome in a randomized study of cesarean skin closure. J Matern Fetal Neonatal Med. 2019 Nov;32(22):3830-3835. doi: 10.1080/14767058.2018.1474870. Epub 2018 May 24. PMID 29739243